CLINICAL TRIAL: NCT07347444
Title: A Prospective, Single-arm, Multicenter, Phase II Clinical Study of Iparomlimab and Tuvoraleimab Injection in Combination With Bevacizumab, Albumin-bound Paclitaxel, and Carboplatin as First- or Second-line Treatment for Patients With Advanced Acral and Mucosal Melanoma
Brief Title: Iparomlimab and Tuvoraleimab Injection in Combination With Bevacizumab, Albumin-bound Paclitaxel, and Carboplatin as First- or Second-line Treatment for Patients With Advanced Acral and Mucosal Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITBAC
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acral Melanoma; Mucosal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvoraleimab injection+Bev+nab-PC (Experimental)
  Interventions: Drug: Iparomlimab and Tuvoraleimab injection+Bev+nab-PC

INTERVENTIONS:
Drug: Iparomlimab and Tuvoraleimab injection+Bev+nab-PC — Iparomlimab and Tuvoraleimab injection: 5mg/kg, D1,Q3W; Bevacizumab: 7.5 mg/kg, D1, Q3W; Albumin-bound paclitaxel: 125mg/m2, D1,8, Q3W; Carboplatin: AUC=2, D1,8, Q3W.

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial designed to evaluate the efficacy and safety of iparomlimab and tuvoraleimab, in combination with bevacizumab, albumin-bound paclitaxel, and carboplatin as first- or second-line treatment in patients with acral and mucosal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (or their legal representatives/guardians) must sign the informed consent form, indicating that they understand the purpose of this study, are aware of the necessary procedures involved, and are willing to participate.
* Aged ≥18 years and ≤75 years, regardless of gender.
* Histologically or pathologically confirmed mucosal or acral melanoma.
* Braf, Nras, and Ckit gene mutation status is unrestricted.
* Unresectable or metastatic melanoma, having received ≤1 prior line of systemic therapy (disease recurrence or metastasis within 6 months after completion of adjuvant therapy is considered as first-line therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 2.
* Expected survival of more than 3 months.
* At least one measurable lesion according to RECIST v1.1. Note: Brain metastases cannot serve as target lesions; Lesions previously treated with radiotherapy cannot serve as target lesions unless imaging demonstrates clear progression.
* Laboratory test results within 7 days prior to screening (including day 7) must meet the following criteria: Neutrophil count ≥1.5×10⁹/L; Platelet count ≥90×10⁹/L; Hemoglobin ≥90 g/L (without transfusion within 14 days); Serum total bilirubin ≤1.25 × upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN (≤5 × ULN for patients with liver metastases); Serum creatinine ≤1.25 × ULN.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose (if the urine pregnancy test result is not conclusively negative, a serum pregnancy test is required, and the serum result shall prevail). If a female subject of childbearing potential engages in sexual activity with a non-sterilized male partner, she must use acceptable contraceptive methods starting from screening and must agree to continue their use for 120 days after the last dose of the study drug; whether to discontinue contraception after this time point should be discussed with the investigator.
* If a non-sterilized male subject engages in sexual activity with a female partner of childbearing potential, he must use effective contraceptive methods from screening until 120 days after the last dose; whether to discontinue contraception after this time point should be discussed with the investigator.
* Subjects are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

* History or presence of other malignancies within the past 5 years, except for cured localized tumors (e.g., basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, etc.).
* Participation in treatment with an investigational drug or use of an investigational device within 4 weeks prior to the first dose of study treatment.
* Palliative local therapy for non-target lesions within 2 weeks prior to the first dose; Non-specific immunomodulatory therapy (e.g., interleukins, interferons, thymosin, etc., excluding IL-11 used for treating thrombocytopenia) within 2 weeks prior to the first dose; Treatment with Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week prior to the first dose.
* Patients who have previously received iparomlimab and tuvoraleimab or other dual immunotherapy, bevacizumab, albumin-bound paclitaxel, or carboplatin.
* Active autoimmune disease that has required systemic treatment in the past two years (i.e., with disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* History of active or documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or chronic diarrhea.
* History of immunodeficiency; Positive HIV antibody test; Current long-term use of systemic corticosteroids or other immunosuppressive agents.
* Known active tuberculosis (TB); Subjects suspected of having active TB must undergo clinical evaluation to rule it out; Known active syphilis infection.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* History of non-infectious pneumonitis/interstitial lung disease that required systemic corticosteroid treatment or current presence of non-infectious pneumonitis.
* Severe infection within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; Active infection requiring systemic anti-infective therapy within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C).
* Subjects with active hepatitis B (HBsAg positive and HBV-DNA >1000 copies/mL [200 IU/mL] or above the lower limit of detection, whichever is higher). Note: Subjects with hepatitis B are required to receive anti-hepatitis B virus therapy during the study treatment.
* Subjects with active hepatitis C (HCV antibody positive and HCV-RNA above the lower limit of detection).
* Major surgical procedure or significant traumatic injury within 30 days prior to the first dose, or planned major surgery within 30 days after the first dose (at the investigator's discretion); Minor local surgery (excluding peripherally inserted central catheter placement and port implantation) within 3 days prior to the first dose.
* Presence of active central nervous system (CNS) metastases; Subjects with previously treated brain metastases are eligible if clinically stable for at least 2 weeks (calculated from the first dose of study drug) and off corticosteroids for at least 3 days prior to the first dose; Subjects with untreated, asymptomatic brain metastases (i.e., no neurological symptoms, no requirement for corticosteroids, and no lesion with longest diameter >1.5 cm) are eligible and require periodic assessment during the study.
* Known brainstem, leptomeningeal, spinal cord metastases, or spinal cord compression.
* Subjects with clinically symptomatic or recurrent pleural effusion, pericardial effusion, or ascites requiring drainage.
* Uncontrolled concurrent illness, including but not limited to symptomatic congestive heart failure (NYHA Class II or higher), unstable angina pectoris, acute myocardial ischemia, poorly controlled arrhythmias, decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the subject's ability to provide written informed consent.
* History of myocarditis, cardiomyopathy, or malignant arrhythmia. Unstable angina, myocardial infarction, congestive heart failure (NYHA Class II or higher), or vascular disease (e.g., aortic aneurysm at risk of rupture) requiring hospitalization within 12 months prior to the first dose, or other cardiac impairment that may affect safety evaluation of the study drug (e.g., poorly controlled arrhythmia, myocardial ischemia); History of esophageal/gastric varices, severe ulcer, unhealed wound, gastrointestinal perforation, abdominal fistula, intra-abdominal abscess, or acute gastrointestinal hemorrhage within 6 months prior to the first dose; Acute exacerbation of chronic obstructive pulmonary disease within 1 month prior to the first dose; Any arterial thromboembolic event, Grade 3 or higher venous thromboembolism per NCI CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to the first dose; Current hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive medication.
* Current significant clinical or imaging evidence of gastrointestinal obstruction.
* History of severe bleeding tendency or coagulation dysfunction; Imaging at screening shows tumor encasement of major blood vessels or significant necrosis/cavitation, and the investigator considers participation may pose a bleeding risk.
* Subjects with tumor invasion of surrounding vital organs or blood vessels (e.g., heart/pericardium, trachea, esophagus, aorta, superior vena cava, etc.), at risk of developing tracheoesophageal fistula, esophagopleural fistula, or enteric fistula, etc.
* Toxicities from prior anti-tumor therapy have not resolved to ≤ Grade 1 per NCI CTCAE v5.0 or to levels specified in the inclusion/exclusion criteria, except for alopecia and residual neuropathy from prior platinum therapy. Subjects with irreversible toxicity not expected to exacerbate with study treatment (e.g., hearing loss) may be included after consultation with the Medical Monitor. Subjects with long-term radiation-induced toxicity judged irreversible by the investigator may be included after consultation with the Medical Monitor.
* Administration of a live vaccine within 30 days prior to the first dose, or planned administration during the study.
* Known allergy to any component of any study drug; History of severe hypersensitivity reaction to other monoclonal antibodies.
* Known history of psychiatric disorder, drug abuse, alcoholism, or substance abuse.
* Pregnant or breastfeeding women.
* Any condition, therapy, laboratory abnormality, or other circumstance that might confound study results, interfere with the subject's participation for the full duration, or participation is not in the best interest of the subject.
* Local or systemic non-malignant disease, or tumor-associated conditions/symptoms that pose significant medical risk and/or uncertainty regarding survival evaluation, such as leukemoid reaction (WBC >20×10⁹/L), cachexia (e.g., known weight loss >10% in the 3 months prior to screening), etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on investigator evaluation.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 2 years
  Defined as the percentage of participants in the analysis population who achieved Complete Response, Partial Response, or Stable Disease, as assessed by the investigator according to RECIST 1.1 criteria.
Duration of Response (DoR) | up to 2 years
  Defined as the time from the first documented confirmed response (CR or PR) to the first documented disease progression (per RECIST 1.1) or death from any cause, whichever occurs first.
Time to Response (TTR) | up to 2 years
  Defined as the time from the first administration of the investigational drug to the first occurrence of Complete Response (CR) or Partial Response (PR).
Progression-Free Survival (PFS) | up to 2 years
  Defined as the time from the initiation of treatment until the first documented disease progression (per RECIST 1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | up to 2 years
  Defined as the time from the initiation of treatment until death from any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university cancer hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No